CLINICAL TRIAL: NCT02832323
Title: Interest of the Peak of Reticulocytes in Chronic Hemodialysis Patients Treated by Mircera
Brief Title: Interest of the Peak of Reticulocytes in Chronic Hemodialysis Patients Treated by Mircera Hemodialysis Population
Acronym: RETICERA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RETICERA
Record Dates: First submitted 2016-06-23; First posted 2016-07-14 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Renal Insufficiency, Chronic
Keywords: hemodialysis; EPO; MIRCERA
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reticera (Other): A blood sample (before dialysis) under the usual conditions will be performed at D0 (= the day of Mircera® injection) and 9 days (+/- 1 day) after each injection Mircera® for hemoglobin and reticulocytes dosage for a period of 6 months.
  Interventions: Biological: Reticera

INTERVENTIONS:
Biological: Reticera — A blood sample (before dialysis) under the usual conditions will be performed at D0 (= the day of Mircera® injection) 9 days (+/- 1 day) after each injection Mircera® for hemoglobin and reticulocytes dosage for a period of 6 months.

SUMMARY:
Patients under hemodialysis treatment are mostly treated by erythropoietin (EPO) through erythropoiesis stimulating agents (ESA). The objective of ESA treatments is to maintain the hemoglobin level in a therapeutic target around 11g/dl. The EPO dose that is necessary to reach this target depends on numerous and imbricated factors such as age, associated pathologies, iron status, inflammation. As of today, there is no marker to predict the EPO response and Hemoglobin (Hb) level is currently the only and late tool to assess the efficacy.

DETAILED DESCRIPTION:
Reticulocytes are immature red blood cells that are temporary present in the blood circulation. They are easily monitored on every automatic dosing machines. Nevertheless, among the dialysis population, they are seldom used and attempt to define a normal reticulocyte level, attesting a correct medullar response to the administrated EPO dose failed due to the timing of blood collection (corresponding to the Nadir day of reticulocytosis).

In a preliminary study, it has shown that reticulocyte count kinetics depends on ESA's type, dose and administration frequency. Reticulocyte kinetics were compared in three groups of stable dialysis patients, depending on their ESA treatment. Reticulocyte curves under a monthly Mircera® treatment were different from the other ESAs, showing a high reticulocyte peak (av. 80 000 reticulocyte/ml) occurring on Day (D)8-D10 after Mircera® administration. On the contrary, at nadir's point (D20-D30 after injection), reticulocyte levels are low for all the patients, preventing from any interpretation of the reticulocyte level at monthly routine assessment. It looks as though it is the peak level of reticulocytes that should be used as a marker of ESA response.

Therefore, monitoring of reticulocytes would support the therapeutic decision on the need to adapt the EPO dose.

The study is design to determinated the interest of the reticulocyte peak in the daily practice

ELIGIBILITY:
Inclusion Criteria:

* Age> or equal to 18 years
* Patients on hemodialysis or hemodiafiltration for at least 3 months
* Patient treated monthly by Mircera® for at least one month
* Affiliate or enjoying a social security scheme
* Patients who received oral and written information about the study, with no objection to the use of personal data and having signed an informed consent form and written

Exclusion Criteria:

* Patient who refused to give his written consent to the study
* Patients treated with another Erythropoiesis stimulating agent
* Minor
* Pregnant or breastfeeding women
* Major under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Reticulocyte peak | Day 9
  variation of the reticulocyte peak compared with hemoglobin level

SECONDARY OUTCOMES:
Mean reticulocyte peak | 6 months
  Reticulocyte peak is collected at D9 after monthly Mircera injection, patient are followed 6 months. The mean of th reticulocyte peak will be calculated at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, PUPH, Principal Investigator — Brest Hospital
Locations (9):
- France (9):
  - CHU Angers, Angers
  - AUB Brest, Brest
  - CHRU La Cavale Blanche, Brest
  - CH Bretagne Sud, Lorient
  - CHRU de Poitiers, Poitiers
  - CH Cornouaille, Quimper
  - CHU Pontchaillou, Rennes
  - CH Yves LE FOLL, Saint-Brieuc
  - Ch Broussais, St-Malo